CLINICAL TRIAL: NCT00851838
Title: Phase 2 Study of Dialysis Efficiency and Tolerability of Peritoneal Dialysis Solution Containing Glucose Plus L-Carnitine in APD (Automated Peritoneal Dialysis) Treated Uremic Patients
Brief Title: L-Carnitine as an Osmo-metabolic Agent for Peritoneal Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-001-06
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2013-03

CONDITIONS: End-Stage Renal Disease
Keywords: Peritoneal dialysis; L-carnitine; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD solution (Experimental)
  Interventions: Drug: L-Carnitine

INTERVENTIONS:
Drug: L-Carnitine — Instillation of glucose-based (1.5 or 2.5 w/v) PD solution containing L-carnitine during the nocturnal exchange in APD treated patients. L-Carnitine (0.1% w/v) is present only in the first 5 Liter APD bag. PD solutions are instilled for 5 days.

SUMMARY:
A major challenge of peritoneal dialysis (PD) therapy is the development of glucose-sparing strategies able to provide an efficacious ultrafiltration (UF) profile. Study hypothesis is to evaluate the possibility to formulate PD solutions containing L-carnitine as an osmotic agent to partially replace glucose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Have a diagnosis of ESRD and have been on Automated Peritoneal Dialysis (glucose 1.5 or 2.5 % w/v) for at least 3 months
* Be in a stable clinical condition during the four weeks immediately prior to Screening Period as demonstrated by medical history, physical examination and laboratory testing
* Have a blood hemoglobin concentration above 8,5 g/100ml (data will be verified with Investigators)
* Have not experienced peritonitis episodes in the last 3 months
* Have Kt/V urea measurement > 1.7 per week in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Have a minimum weekly creatinine clearance of 45 litres in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Have a D/P Creatinine ratio at Peritoneal Equilibration Test (PET) between 0.50 and 0.81 in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Have a D/P Glucose ratio at Peritoneal Equilibration Test (PET) between 0.26 and 0.49 in a previous test performed within 6 months that should be confirmed at Baseline Visit
* Be treated by the participating clinical Investigator for a period of at least three months
* Have understood and signed the Informed Consent Form.

Exclusion Criteria:

* Have a history of drug or alcohol abuse in the six months prior to entering the protocol
* Be in treatment with androgens
* Have Diabetes Mellitus (as defined by the American Diabetes Society, objectively documented by a fasting plasma glucose and HbA1c determinations)
* Have clinically significant abnormal liver function test (SGOT, SGPT, and gamma-GT > 2 times the upper normal limit)
* Have acute infectious conditions (i.e.: pulmonary infection, acute hepatitis, high or low urinary tract infections, renal parenchymal infection, pericarditis, etc)
* Have a history of congestive heart failure and clinically significant arrhythmia
* Have an history of epilepsy or any NCS disease
* Have malignancy within the past 5 years, including lymphoproliferative disorders
* Have any medical condition that, in the judgment of the Investigator, would jeopardize the patient's safety following exposure to study drug, particularly if patient's life expectancy is less than 1 year
* Have a history of L-Carnitine therapy or use in the month prior to entering the protocol
* Have used any investigational drug in the 3 months prior to entering the protocol
* Be in pregnancy, lactation, fertility age without protection against pregnancy by adequate contraceptive means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of L-Carnitine containing PD solution on peritoneal ultrafiltration | day 5

CONTACTS AND LOCATIONS:
Overall Officials: Mario Bonomini, MD, Principal Investigator — G. d'Annunzio University; Arduino Arduini, MD, Study Director — Iperboreal Pharma Srl
Locations (1):
- Division of Nephrology, University of "G. d'Annunzio", Chieti, Italy